CLINICAL TRIAL: NCT04718337
Title: Postpartum Intra-caesarean Intrauterine Device Insertion Using a Novel Technique
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Christine Tamer Laisha, Doctor, Assiut University
Other Study IDs: Postpartum IUD insertion
Record Dates: First submitted 2020-09-26; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: IUD Complication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The assessment of efficacy and patient safety of immediate postpartum IUD insertion using a novel technique.

DETAILED DESCRIPTION:
The postpartum period is so critical time for both the mother and newborn that needs special health care because there are high morbidity and mortality rates during it (1).

The World Health Organization (WHO) recommends that a woman should wait at least 24 months after delivery before the next pregnancy to decrease the adverse maternal, perinatal ,and infant outcomes (2, 3).

A woman's fertility may begin to return rapidly and ovulate within 4:6 weeks postpartum particularly if she is not exclusively breastfeeding. In addition , more than 50% of women become sexually active by 6 weeks postpartum (4, 5).

So, it is important to provide highly effective contraception immediately after delivery before leaving the delivery setting especially in communities where women cannot return easily for follow up visits due to financial and social barriers or who have limited access to medical service (6, 7).

The use of effective postpartum contraception particularly longـacting reversible contraception (LARC) methods like the intrauterine device (IUD) has been shown to decrease the risk of unintended pregnancy and its complications and avoid repeated caesarean sections with higher continuation rates of use than other methods 6 months after delivery (8-10).

Immediate post placental intraـcaesarean IUD insertion has many advantages as it is effective reversible longـterm contraception, doesn't interfere with breastfeeding, is coitus independent and the woman can avoid discomfort and pain during the standard insertion and bleeding from insertion will be masked by lochia (11-14).

Studies have shown that with effective provider training, the immediate postpartum IUD insertion (IPPIUD) complications such as expulsion, pelvic infection, bleeding, pain, missing threads ,and failure rates are not significantly different from those of interval PPIUD insertion (4:6 weeks) after delivery (15, 16).

By using a novel technique in this study, these complications would be decreased.

ELIGIBILITY:
Inclusion Criteria:

1. Women admitted to undergo CS.
2. Singleton pregnancy.
3. Delivery of a liveـborn infant with gestational age < 36 weeks.
4. Informed and written consent to participate in the study.

Exclusion Criteria:

1. History of dysmenorrhea, menorrhagia or coagulopathies.
2. Uterine anomalies or fibroids.
3. Antepartum or intrapartum hemorrhage.
4. Prolonged rupture of membranes <24 hours with or without chorioamnionitis.
5. Intrapartum fever.
6. History of current, recent (within previous 3 months) or recurrent pelvic infilammatory diseases (PID).
7. History of ectopic pregnancy.
8. Multiple pregnancy.
9. Active cervicitis, vaginitis or sexual transmitted diseases (STD) on gyaecological examination.
10. Allergy to any component of the IUD or Wilson's disease.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy of postpartum intra-caesaren IUD insertion | 6 months
  the evaluation of efficacy of this novel technique to decrease the rates of expulsion, missing threads and failure.

SECONDARY OUTCOMES:
Patient safety of postpartum intra-caesarean IUD insertion | 6 months
  the evaluation of patient safety including pelvic infections, lower abdominal pain and excessive bleeding.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kumar M, Kumar M, Aggarwal P, Gangania A, Dewan. A study to evaluate and compare the expulsion and continuation rates of post placental insertion of Cu 375 and CuT 380A in Indian women at a premier hospital in New Delhi, India. Int J Reprod Contracept Obstet Gynecol 2017;6(9):3992-4000. Health WHODoM, Abuse S, Organization WH, Health WHODoM, Health SAM, Evidence WHOMH, et al. Mental health atlas 2005: World Health Organization; 2005. Rutstein S, Johnson K, Conde-Agudelo A, Rosas-Bermudez A. Effect of birth spacing on infant and child mortality: a systematic review and meta-analysis. WHO Technical Consultation and Scientific Review of Birth Spacing 2005;13(5). Jackson E, Glasier A. Return of ovulation and menses in postpartum nonlactating women: a systematic review. Obstet Gynecol 2011;117(3):657-662. Speroff L, Mishell DR. The postpartum visit: it's time for a change in order to optimally initiate contraception. Contraception 2008;78(2):90-98. Lucksom PG, Kanungo BK, Sebastian N, Mehrotra R, Pradhan D, Upadhya R. Comparative study of interval versus postpartum Cu-T insertion in a central referral hospital of North East India. Int J Reprod Contracept Obstet Gynecol 2015;4(1):47-51. DiBari JN, Yu SM, Chao SM, Lu MC. Use of postpartum care: predictors and barriers. Journal of pregnancy 2014;2014. Levi EE, Stuart GS, Zerden ML, Garrett JM, Bryant AG. Intrauterine device placement during cesarean delivery and continued use 6 months postpartum: a randomized controlled trial. Obstet Gynecol 2015;126(1):5-11. Organization WH. Report of a WHO technical consultation on birth spacing: Geneva, Switzerland 13-15 June 2005. World Health Organization; 2007. Obstetricians ACo, Obstetrics GJ, gynecology. ACOG Practice Bulletin No. 121: Long-acting reversible contraception: Implants and intrauterine devices. Obstetrics and Gynecology. 2011;118(1):184-196. Kapp N, Curtis KM. Intrauterine device insertion during the postpartum period: a systematic review. Contraception 2009;80(4):327-336. Glasier A. Best Practice in Postpartum Family Planning. Best Practice Paper No 1. June 2015. London: Royal College of Obstetricians and Gynaecologists; 2015. Heller R, Cameron S, Briggs R, Forson N, Glasier A. Postpartum contraception: a missed opportunity to prevent unintended pregnancy and short inter-pregnancy intervals. J Fam Plann Reprod Health Care 2016;42(2):93-98. Teal SB. Postpartum contraception: optimizing interpregnancy intervals. Contraception 2014;89(6):487-488. Grimes DA, Lopez LM, Schulz KF, Van Vliet HA, Stanwood NL. Immediate post-partum insertion of intrauterine devices. Cochrane Database Syst Rev 2010;(5):CD003036. Çelen Ş, Sucak A, Yıldız Y, Danışman N. Immediate postplacental insertion of an intrauterine contraceptive device during cesarean section. Contraception 2011;84(3):240-243. Zaconeta AM, Oliveira AC, Estrela FS, Vasconcelos TM, França PS, Wanderley MdS, Amato AA. Intrauterine device insertion during cesarean section in women without prenatal contraception counseling: lessons from a country with high cesarean rates. Revista Brasileira de Ginecolgia e Obstetricia 2019;41(8):485-492.